CLINICAL TRIAL: NCT05084560
Title: Development of AWZ1066S, a Small Molecule Anti-Wolbachia Candidate Macrofilaricide Drug
Acronym: AWOL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety issues
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government); Covance (Industry); Subiaco Associates Limited (Unknown); Sylexis Limited (Unknown); Eisai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-059
Record Dates: First submitted 2021-10-05; First posted 2021-10-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Filariasis, Lymphatic; Onchocerciasis
Keywords: Lymphatic filariasis; Onchocerciasis; Wolbachia; Phase 1; Healthy volunteers; Randomized; Double blind; Placebo
MeSH Terms: conditions — Elephantiasis, Filarial; Onchocerciasis

STUDY DESIGN:
Intervention Model Description: Sequential, ascending dose design, double-blind, placebo controlled.
  Part A: single ascending dose design with 6 dosing levels. Part B: multiple ascending dose design with 4 dosing levels.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AWZ1066S (Experimental): AWZ1066S
  Part A Cohort A1- 100mg single dose Cohort A2- 200mg single dose Cohort A3- 400mg single dose Cohort A4- 800mg fasted single dose and 800mg fed single dose Cohort A5- 1200mg single dose Cohort A6- 1600mg single dose
  The doses for part B will be selected following review of data from Part A. Cohort B1- AWZ1066S once daily for 7 days Cohort B2- AWZ1066S once daily for 7 days Cohort B3- AWZ1066S once daily for 7 days Cohort B4- AWZ1066S once daily for 7 days
  Interventions: Drug: AWZ1066S
- Placebo (Placebo Comparator): Placebo
  Cohort A1- equivalent placebo single dose Cohort A2- equivalent placebo single dose Cohort A3- equivalent placebo single dose Cohort A4- equivalent placebo fasted single dose and equivalent placebo fed single dose Cohort A5- equivalent placebo single dose Cohort A6- equivalent placebo single dose
  The doses for part B will be selected following review of data from Part A. Cohort B1- equivalent placebo once daily for 7 days Cohort B2- equivalent placebo once daily for 7 days Cohort B3- equivalent placebo once daily for 7 days Cohort B4- equivalent placebo once daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AWZ1066S — Candidate drug to treat lymphatic filariasis by targeting Wolbachia endosymbiont
  Arms: AWZ1066S
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Lymphatic filariasis and onchocerciasis are a group of neglected tropical diseases caused by the transmission of worm larvae (microfilaria) by biting insects. Once a human is infected, the larvae mature into adult worms that release huge numbers of larvae into the lymphatics for 5-15 years. The larvae cause tissue damage resulting in the disabling diseases of elephantiasis (gross leg and scrotal swelling) and river blindness. These diseases affect 160 million people and are acknowledged major public health problems in the tropics. Current treatments mainly target the larvae but not the adult worms that live for years, meaning that repeated courses of treatment over many years are needed. These repeated courses are usually delivered at population level in the form of mass drug administration programmes.

For the adult worms to be able to grow, reproduce and infect more humans they are dependent on a bacterium which lives inside them. This bacterium (Wolbachia) is not naturally found in humans. Some drugs are able to target Wolbachia, however they are unsuitable for mass drug administration programmes because they have to be given for 4-6 weeks and cannot be used in children or pregnant women.

AWZ1066S is a novel drug developed in Liverpool that has been shown in experimental models to target Wolbachia and indirectly kill the adult parasitic worms after a 7 day course. After extensive safety testing in animals we are conducting a Phase 1, first in human study, to assess the safety, tolerability and pharmacokinetics of ascending single and multiple oral doses of AWZ1066S in healthy volunteers. The study is a single centre study, will last approximately 1 year and will take place in a dedicated Phase 1 trial unit. Depending on which group they are enrolled into, participants will take either one dose, two doses or seven doses and their involvement will last between 38 and 45 days. Participants will be closely monitored for adverse effects.

DETAILED DESCRIPTION:
AWZ1066S is in the early stages of clinical development, for safety reasons, a sequential, ascending dose design is being used. The study is double-blind, and placebo controlled. All research activities will be conducted within a dedicated Phase 1 Clinical Research Facility.

Part A comprises a single ascending dose design with an overall group total of 48 participants. These will be studied in 6 cohorts (Cohorts A1 to A6), with each cohort consisting of 8 participants (6 randomised to oral dose of AWZ1066S and 2 randomised to placebo). Each participant will receive single dose of AWZ1066S, apart from cohort A4 participants who will take a single dose when fasting and and a single dose when fed, separated by a minimum of 7 days.

The planned doses for Part A are:

Cohort A1- 100mg Cohort A2- 200mg Cohort A3- 400mg Cohort A4- 800mg fasted and 800mg fed Cohort A5- 1200mg Cohort A6- 1600mg Participants will receive their dose whilst resident in the Clinical Research Facility and will return for outpatient visits on Day 3, 4 and 10 safety assessments and pharmacokinetic blood samples.

Part B comprises a multiple ascending dose design, to investigate 4 dose levels in four cohorts (cohorts B1 to B4) with each cohort consisting of 8 participants (6 randomised to oral dose of AWZ1066S and 2 randomized to placebo). The doses investigated will be selected following review of data from the single dosing study (Part A). The intention is to enrol a minimum 32 healthy participants. Each participant will receive single daily dose of AWZ1066S for 7 days. Participants will receive their dose whilst resident in the Clinical Research Facility and will return for outpatient visits on Day 3, 5, 9 and 10 for safety assessments and pharmacokinetic blood samples. A second resident period on Day 6 to Day 8 will allow pharmacokinetic blood samples and safety assessments.

Safety and tolerability will be monitored by adverse events, vital signs, ECGs, urinalysis, routine haematology and biochemistry. Escalation of dosing will only take place after examination of safety data by the Dose Escalation Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants 2 aged 18-65 years 3 BMI 18.0-35.0 kg/m2, maximum weight 100 kg 4 in good health, as determined by: 4a medical history, 4b physical examination, 4c vital signs assessment, 4d 12-lead ECG 4e clinical laboratory evaluations 5 provision of informed consent and abide by study restrictions

Exclusion Criteria:

1. not willing to abide by contraception restrictions
2. donated blood in previous 3 months, plasma previous 7 days, platelets previous 6 weeks
3. consumption >14 units of alcohol/week
4. tobacco smoking
5. concomitant medication, apart from treatments for mild asthma, eczema, contraception, paracetamol
6. herbal remedies
7. history of anaphylaxis, drug allergy, clinically significant atopic condition as determined by Investigator
8. clinically significant medical history, as determined by the Investigator
9. positive hepatitis, HIV serology
10. live vaccine in previous 3 months, Covid-19 vaccine prior 14 days
11. Participants who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | From day of first dose to 10 days after last dose
  Number

SECONDARY OUTCOMES:
Single dose pharmacokinetics Cmax | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, maximum plasma concentration (Cmax)
Single dose pharmacokinetics tmax | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, time to reach maximum plasma concentration (tmax)
Single dose pharmacokinetics t1/2 | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, half life (t1/2)
Single dose pharmacokinetics CL/F | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, apparent total clearance after oral administration (CL/F)
Multiple dose pharmacokinetics Cmax | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, maximum plasma concentration (Cmax)
Multiple dose pharmacokinetics tmax | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, time to reach maximum plasma concentration (tmax)
Multiple dose pharmacokinetics t1/2 | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, half life (t1/2)
Multiple dose pharmacokinetics CL/f | From day of first dose to 10 days after last dose
  Pharmacokinetic parameter, apparent total clearance after oral administration (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Devereux, MD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Commercial sensitivity

REFERENCES:
- [Background] Hong WD, Benayoud F, Nixon GL, Ford L, Johnston KL, Clare RH, Cassidy A, Cook DAN, Siu A, Shiotani M, Webborn PJH, Kavanagh S, Aljayyoussi G, Murphy E, Steven A, Archer J, Struever D, Frohberger SJ, Ehrens A, Hubner MP, Hoerauf A, Roberts AP, Hubbard ATM, Tate EW, Serwa RA, Leung SC, Qie L, Berry NG, Gusovsky F, Hemingway J, Turner JD, Taylor MJ, Ward SA, O'Neill PM. AWZ1066S, a highly specific anti-Wolbachia drug candidate for a short-course treatment of filariasis. Proc Natl Acad Sci U S A. 2019 Jan 22;116(4):1414-1419. doi: 10.1073/pnas.1816585116. Epub 2019 Jan 7. PMID 30617067